CLINICAL TRIAL: NCT06926998
Title: An Open-Label, Multicenter Phase Ib/ll Clinical Study Evaluating the Safety and Efficacy of 9MW2821 Combined With Other Antitumor Drugs in Patients With Advanced Gynecological Tumors
Brief Title: 9MW2821 Combined With Other Antitumor Drugs in Patients With Advanced Gynecological Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9MW2821-CP204
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Gynecological Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental): 9MW2821+ other anti-cancer therapy
  Interventions: Drug: 9MW2821+other anticancer therapy

INTERVENTIONS:
Drug: 9MW2821+other anticancer therapy — Subjects will receive intravenous (IV) infusion of 9MW2821 +other anticancer therapy as per protocol

SUMMARY:
To evaluate the safety, tolerability, and preliminary efficacy of 9MW2821 in combination with other anti-tumor agents in patients with advanced gynecological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Competent to comprehend, sign, and date an independent ethics committee/institutional review board/research ethics board (IEC/IRB/REB) approved informed consent form.
2. Female subjects aged 18 to 75 years (including 18 and 75 years).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histopathological diagnosed of advanced gynecological tumors.
5. Subjects must submit tumor tissues for test.
6. Life expectancy of ≥ 12 weeks.
7. Subjects must have measurable disease according to RECIST (version 1.1).
8. Adequate organ functions.
9. Sexually active fertile subjects must agree to use methods of contraception during the study and at least 180 days after termination of study therapy.
10. Subjects are willing to follow study procedures.

Exclusion Criteria:

1. History of another malignancy within 3 years before the first dose of study drug.
2. Patients with ongoing clinically significant toxicities related to prior treatment.
3. Presence of Grade ≥ 2 peripheral neuropathy.
4. Exclusion of prior diseases and prior treatments as specified in the protocol.
5. Comorbidities: a. Hemoglobin A1C ≥ 8%; b. Ocular diseases or symptoms present prior to the first dose of study medication; c. Severe respiratory diseases; d. Clinically significant cardiovascular or cerebrovascular diseases within 6 months prior to the first dose of study medication; e. Active autoimmune diseases within 2 years prior to the first dose of study medication, or a history of autoimmune diseases with potential for recurrence; f. Active infections; g. Severe arterial or venous thromboembolic events.
6. Clinically significant bleeding symptoms or a clear bleeding tendency within 3 months prior to the first dose of medication.
7. Subjects with central nervous system (CNS) metastases and/or carcinomatous meningitis.
8. Pleural, peritoneal, or pericardial effusion with clinical symptoms or requiring repeated drainage procedures.
9. Prior Treatments: a. Major surgical procedures within 28 days prior to the first dose of study medication; b. Administration of other investigational drugs or experimental medical devices within 28 days prior to the first dose of study medication; c. Use of P-glycoprotein inhibitors or inducers, or potent CYP3A4 inhibitors within 14 days prior to the first dose of study medication; d. Receipt of live vaccines within 28 days prior to the first dose of study medication or planned administration of any live vaccine during the study period; e. Prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation;.
10. Subjects with a history of drug abuse or psychiatric disorders, or suspected allergy, intolerance, or severe infusion reactions to the investigational drug or any of its components.
11. Pregnant or lactating women.
12. Not suitable to receive study treatment for other conditions as per investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 24 months
  Objective Response Rate

SECONDARY OUTCOMES:
DoR | Up to 24 months
  Duration of Response
TTR | Up to 24 months
  Time to Response
DCR | Up to 24 months
  Disease Control Rate
PFS | Up to 24 months
  Progression Free Survival
OS | Up to 24 months
  Overall Survival
Pharmacokinetic parameter：total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) | 24 months
  Maximum observed concentration (Cmax)
Pharmacokinetic parameter：total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) | 24 months
  Area under the concentration-time curve (AUC)
Pharmacokinetic parameter：total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) | 24 months
  Half-life (t1/2)
Pharmacokinetic parameter：total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) | 24 months
  Clearance (CL)
Incidence of Anti-Drug Antibody (ADA) | 24 months
  ADA

CONTACTS AND LOCATIONS:
Overall Officials: Hanmei Lou, Professor, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No